CLINICAL TRIAL: NCT02865213
Title: Assessment of Skeletal and Dentoalveolar Changes Resulting From Posterior Teeth Intrusion in Treatment of the Anterior Open Bite - a Randomized Controlled Trial
Brief Title: Molar Intrusion in Open Bite Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-01-2016
Record Dates: First submitted 2016-07-22; First posted 2016-08-12 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Anterior Open Bite
Keywords: Open bite; Molar intrusion; Temporary anchorage devices
MeSH Terms: conditions — Open Bite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Miniplates + OBA (Experimental): The intrusion of posterior teeth using Miniplates + OBA will be performed. The investigators will apply a modified version of the OBA (Open Bite Appliance), by Erverdi and Usumez, for all patients in upper posterior teeth and miniplates.
  The miniplates are for Jeil Dual top® anchor system, Jeil medical corporation, #702,kolon science valley 2nd, 811, Guro-Dong, Guro-Gu, Seoul, 152-050, Korea. Tel: 82.2.850.3500. Fax: 82.2.850.3537. homepage: www.jeilmed.co.kr/ E-mail: mktg@jeilmed.co.kr
  Interventions: Device: OBA; Device: Miniplates
- Miniscrews + OBA (Experimental): The intrusion of posterior teeth using Miniscrews + OBA will be performed. The investigators will apply a modified version of the OBA (Open Bite Appliance), by Erverdi and Usumez, for all patients in upper posterior teeth and miniscrews.
  The miniscrews are for Denxy ® dental orthodontic products, Denxy technology co, limited . 404,Lihuabuilding,Furongroad, Changsha, Hunan, China. Tel: 0086-731-89717339. Fax: 0086-731-82237315. Homepage: www.denxy-orthodontic.com/email: DENXYDENTALBOSS@126.COM
  Interventions: Device: OBA; Device: Miniscrews
- Only OBA (Experimental): The intrusion of posterior teeth using OBA only will be performed. The investigators will apply a modified version of the OBA (Open Bite Appliance), by Erverdi and Usumez, for all patients in upper posterior teeth only.
  Interventions: Device: OBA

INTERVENTIONS:
Device: OBA — The intrusion of posterior teeth using removable appliance "OBA".
Device: Miniplates — The intrusion of posterior teeth using temporary anchorage "Miniplates".
  Arms: Miniplates + OBA
Device: Miniscrews — The intrusion of posterior teeth using temporary anchorage "Miniscrews".
  Arms: Miniscrews + OBA

SUMMARY:
This experimental study will evaluate the effect of different methods for the molar intrusion (compared with the control group) in adolescent and adult patients with open bite malocclusion. The study sample will consist of 45 patients with anterior open bite. The sample will be randomly allocated into two experimental groups, in addition to a control group.

The investigators will apply a modified version of the Open Bite Appliance (OBA), by Erverdi and Usumez, for all patients in upper posterior teeth. For this purpose, miniplates will be used in the first treatment group, while miniscrews will be used in the second treatment group. In the control group, only OBA will be used. The skeletal and dentoalveolar changes occurring after intrusion of posterior teeth will be assessed by using posteroanterior and lateral cephalometric radiographs. Pre- and post- treatment changes for each group will be evaluated, in addition to the comparison of the post-treatment skeletal and dental changes that occurs between groups.

DETAILED DESCRIPTION:
Open bite malocclusion is considered one of the most difficult orthodontic problems to correct because it appears as a result of the interaction of numerous etiological factors (genetic, dental, skeletal, functional, soft tissue, and habit) that contribute to its development. Various therapeutic approaches have been proposed for the treatment of an anterior open bite. These approaches vary depending on the causative factors and involve myotherapy, preventive treatment, functional therapy, orthognathic surgery, and orthodontic treatment using anterior teeth extrusion or posterior teeth intrusion. Among the non-surgical orthodontic treatment methods are the temporary anchorage devices (TADs) including miniplates and miniscrew or micro-screw implants. The intrusion of posterior teeth with temporary anchorage devices was suggested to lead to decreased lower facial height by a counterclockwise rotation of the mandible; this may resemble the orthognathic surgery outcomes for any open bite patients. To the best of the investigators current knowledge, this is the first randomized controlled trial evaluating the effect of molar intrusion in adolescence and adult patients in the permanent dentition stage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with skeletal open bite determined by an increased B angle (angle between the maxillary plane and mandibular plane), the Sum of Bjork and the mandibular plane angle (angle between SN plane and mandibular plane).
* Patients between 12 and 18 years old in permanent dentition stage.
* Negative over-bite of more than a mm
* Class I or Class II skeletal anteroposterior relationship.

Exclusion Criteria:

* Previous orthodontic treatment.
* Patients with syndromes, clefts, or craniofacial abnormalities.
* Class III skeletal anteroposterior relationship.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Overbite | This variable will be evaluated twice; T0 before treatment, and T1 at the end of molar intrusion which will be approximately after 7 months
  The distance between the incisal edges of upper incisors and the incisal edges of the lower incisors, measured in mm

SECONDARY OUTCOMES:
Molar intrusion | This variable will be evaluated twice; T0 before treatment, and T1 at the end of molar intrusion which will be approximately after 7 months
  The vertical distance between upper molars and the true horizontal plane (measured in mm).
Mandibular autorotation | This variable will be evaluated twice; T0 before treatment, and T1 at the end of molar intrusion which will be approximately after 7 months
  This variable will be measured by superimposition of the anterior cranial base.
Anterior facial height | This variable will be evaluated twice; T0 before treatment, and T1 at the end of molar intrusion which will be approximately after 7 months
  The distance between the point "N" and the point "Me"
Change in the anteroposterior position of the point "B" | This variable will be evaluated twice; T0 before treatment, and T1 at the end of molar intrusion which will be approximately after 7 months
  The horizontal distance between point "B" and the true vertical plane.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Yousef, DDS MSc PhD, Study Chair — Damascus University
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No
No
  Individual participant data will be only available to the researchers in the department of Orthodontics, Damascus University

REFERENCES:
- [Background] Ng J, Major PW, Flores-Mir C. True molar intrusion attained during orthodontic treatment: a systematic review. Am J Orthod Dentofacial Orthop. 2006 Dec;130(6):709-14. doi: 10.1016/j.ajodo.2005.05.049. PMID 17169732
- [Background] Sugawara J, Baik UB, Umemori M, Takahashi I, Nagasaka H, Kawamura H, Mitani H. Treatment and posttreatment dentoalveolar changes following intrusion of mandibular molars with application of a skeletal anchorage system (SAS) for open bite correction. Int J Adult Orthodon Orthognath Surg. 2002;17(4):243-53. PMID 12592995
- [Background] Deguchi T, Kurosaka H, Oikawa H, Kuroda S, Takahashi I, Yamashiro T, Takano-Yamamoto T. Comparison of orthodontic treatment outcomes in adults with skeletal open bite between conventional edgewise treatment and implant-anchored orthodontics. Am J Orthod Dentofacial Orthop. 2011 Apr;139(4 Suppl):S60-8. doi: 10.1016/j.ajodo.2009.04.029. PMID 21435540
- [Background] Akan S, Kocadereli I, Aktas A, Tasar F. Effects of maxillary molar intrusion with zygomatic anchorage on the stomatognathic system in anterior open bite patients. Eur J Orthod. 2013 Feb;35(1):93-102. doi: 10.1093/ejo/cjr081. Epub 2011 Aug 9. PMID 21828357
- [Background] Xun C, Zeng X, Wang X. Microscrew anchorage in skeletal anterior open-bite treatment. Angle Orthod. 2007 Jan;77(1):47-56. doi: 10.2319/010906-14R.1. PMID 17029531
- [Background] Erverdi N, Keles A, Nanda R. The use of skeletal anchorage in open bite treatment: a cephalometric evaluation. Angle Orthod. 2004 Jun;74(3):381-90. doi: 10.1043/0003-3219(2004)0742.0.CO;2. PMID 15264651
- [Background] Hart TR, Cousley RR, Fishman LS, Tallents RH. Dentoskeletal changes following mini-implant molar intrusion in anterior open bite patients. Angle Orthod. 2015 Nov;85(6):941-8. doi: 10.2319/090514-625.1. Epub 2014 Dec 22. PMID 25531420
- [Background] Kuroda S, Katayama A, Takano-Yamamoto T. Severe anterior open-bite case treated using titanium screw anchorage. Angle Orthod. 2004 Aug;74(4):558-67. doi: 10.1043/0003-3219(2004)0742.0.CO;2. PMID 15387036